CLINICAL TRIAL: NCT02070536
Title: Predictive Values of Plasma Soluble RAGE Levels and RAGE Polymorphisms for the Onset of Acute Respiratory Distress Syndrome in Critically Ill Patients
Acronym: PrediRAGE
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0182
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2014-02

CONDITIONS: Intensive Care Unit; Population at High Risk for ARDS Development
Keywords: Acute Respiratory Distress Syndrome (ARDS); Receptor for advanced glycation end products (RAGE); Soluble RAGE (sRAGE); Gene polymorphisms; Biomarker
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ARDS (Acute Respiratory Distress Syndrome)
  Interventions: Other: sRAGE

INTERVENTIONS:
Other: sRAGE

SUMMARY:
Current clinical prediction scores for acute respiratory distress syndrome (ARDS) have limited positive predictive value. No studies have evaluated predictive kinetics of plasma biomarkers and receptor for advanced glycation end products (RAGE) polymorphisms in a broad population of critically ill patients or as an adjunct to clinical prediction scores.

The main objective of the investigators study is to evaluate the predictive values of plasma soluble RAGE levels for the onset of ARDS in a high risk population of patients admitted to the intensive care unit (ICU).

One of the investigators goals is to improve early identification of patients at risk for ARDS in order to better implement preventive stategies prior to ARDS development.

The primary outcome is the occurrence of ARDS during the first week after admission to the ICU.

DETAILED DESCRIPTION:
BACKGROUND :

ARDS is a major cause of morbidity and mortality in critically ill patients. Only few pharmacological treatments are available, with limited evidence of efficacy.

The development of efficient preventive stategies is limited by the investigators inability to predict which patients are likely to develop ARDS. The Lung Injury predicition Score (LIPS) has been developed to identify patients at high risk for ARDS, but its predictive value remains limited.

The receptor for advanced glycation end product (RAGE) is now identified as a marker of alveolar type I cell injury. RAGE is a member of the immunoglobulin superfamily that acts as a multiligand receptor which is involved in propagating inflammatory responses. Plasma levels of sRAGE are correlated with clinical and radiologic severity in ARDS patients.

The investigators main objective is to assess the predictive values of plasma sRAGE and esRAGE levels, as well as their evolution over the first 24 hours after admission, for the onset of ARDS in high risk patients.

The secondary objectives are to :

* to evaluate the predictive value of RAGE polymorphisms (_429 T/C, _374 T/A, 2184 A/G, Gly82Ser) for the onset of ARDS
* to evaluate the predictive value of maximal plasma levels of RAGE soluble forms for the onset of ARDS
* to test the relationship between RAGE polymorphisms and plasma sRAGE and esRAGE levels
* to test whether serial sRAGE measurements would improve the discrimination of the LIP Score or not
* to evaluate the prognostic value of plasma levels of RAGE soluble forms for : duration of mechanical ventilation, length of stay in the ICU and 30-day mortality.

DESIGN NARRATIVE :

The purpose of this prospective observational study is to test the values of RAGE polymorphism and soluble forms plasma levels for ARDS prediction in high risk ICU patients

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU
* Patients presenting with risk factors for ARDS : high risk surgery, sepsis, shock, panceatitis, pneumonia, aspiration, drowning, massive transfusion, pulmonary contusion, serious burn, severe trauma.
* Informed consent

Exclusion Criteria:

* Pregnancy
* Age < 18 years
* Criteria for ARDS at admission to the ICU
* Expected survival under 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population at high risk for ARDS development
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
development of ARDS | during the first week after admission to the ICU
  The development of ARDS, based on Berlin definition criteria, during the first week after admission to the ICU

SECONDARY OUTCOMES:
Plasma sRAGE and esRAGE levels | at ICU admission (Day 0)
Plasma sRAGE and esRAGE levels | (Day 1)
Evolution of plasma sRAGE levels | between day 0 and day 1
Maximal plasma levels of sRAGE and esRAGE | during the first 24 hours after ICU admission
Development of ARDS | during at day 14 and day 30 after ICU admission
Total duration of mechanical ventilation | at day 1
Length of stay in ICU | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu JABAUDON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Blondonnet R, Joubert E, Godet T, Berthelin P, Pranal T, Roszyk L, Chabanne R, Eisenmann N, Lautrette A, Belville C, Cayot S, Gillart T, Souweine B, Bouvier D, Blanchon L, Sapin V, Pereira B, Constantin JM, Jabaudon M. Driving pressure and acute respiratory distress syndrome in critically ill patients. Respirology. 2019 Feb;24(2):137-145. doi: 10.1111/resp.13394. Epub 2018 Sep 5. PMID 30183115
- [Derived] Pranal T, Pereira B, Berthelin P, Roszyk L, Godet T, Chabanne R, Eisenmann N, Lautrette A, Belville C, Blondonnet R, Cayot S, Gillart T, Skrzypczak Y, Souweine B, Bouvier D, Blanchon L, Sapin V, Constantin JM, Jabaudon M. Clinical and Biological Predictors of Plasma Levels of Soluble RAGE in Critically Ill Patients: Secondary Analysis of a Prospective Multicenter Observational Study. Dis Markers. 2018 May 10;2018:7849675. doi: 10.1155/2018/7849675. eCollection 2018. PMID 29861796